CLINICAL TRIAL: NCT04404257
Title: Reduce Radiation Exposure in Fluoroscopic Interventions Evaluation (REDEFINE): A Prospective, Randomized Evaluation of the ControlRad System to Reduce Radiation Exposure During Cardiac Catheterization and Electrophysiology (EP) Procedures.
Brief Title: Reduce Radiation Exposure in Fluoroscopic Interventions Evaluation
Acronym: REDEFINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Simon Dixon, MD, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-174
Record Dates: First submitted 2020-04-08; First posted 2020-05-27 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Cardiac Catheterization; Radiation Exposure
Keywords: ControlRad System; Cardiac Catheterization; Radiation Exposure; Fluoroscopic x-ray

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 like a flip of a coin, to receive either cardiac catheterization and or electrophysiology implant procedures without ControlRad system or cardiac catheterization and or electrophysiology (EP) implant procedures with the ControlRad system.
Who Masked: Participant
Masking Description: Participant will be blinded to the arm assigned to; but the investigators, cath lab operators and staff will be informed of the randomized assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- ControlRad System (Experimental): Participant will undergo Cardiac catheterization or electrophysiology implant procedures with the ControlRad system installed in Cath lab room 5
  Interventions: Radiation: ControlRad System
- Without ControlRad System (Active Comparator): Participant will undergo the cardiac catheterization or electrophysiology implant procedures per standard of care. Meaning, without the ControlRad system installed in Cath lab room 5.
  Interventions: Radiation: Without ControlRad System

INTERVENTIONS:
Radiation: ControlRad System — Cardiac Catheterization or electrophysiology implant procedures with Control Rad system device installed in the cath lab room #5.
  Arms: ControlRad System
Radiation: Without ControlRad System — Cardiac Catheterization or electrophysiology implant procedures in cath lab room 5 without the ControlRad system device.
  Arms: Without ControlRad System

SUMMARY:
The purpose of this study is to determine whether the ControlRad system device when installed in Fluoroscopic (x-ray) machine reduces radiation dose to operators (Doctors and nurses) and to the patient who is undergoing cardiac Catheterization and electrophysiology (EP) implant procedures.

DETAILED DESCRIPTION:
This is a Prospective, randomized (like a "flip of a coin") single center study evaluating the ControlRad system device when installed - retrofitted on existing C-arms for fluoroscopy (x-ray) will reduce radiation exposure without compromising image quality in the region of interest and overall workflow during cardiac catheterization and electrophysiology (EP) implant procedures. Enrollment will be limited to 40 cardiac catheterization, and 30 pacemaker and/or ICD procedures. All patients presenting to Beaumont Hospital Royal Oak who are scheduled for cardiac catheterization with coronary angiography and electrophysiology implant in Cath Lab 5 where device is installed will be considered for inclusion in the study. Physicians and staff (20 fellows; 35 attending physicians; and 56 Cath-lab staff,including Nurse/Anesthesia team) will be invited to participate in the study. For each procedure, 3 staff members will be study subjects: a) the primary operator, b) the secondary operator, c) the nurse/tech and or Anesthetist who circulates in the room. Different operators and staff may participate in each case depending on cath-lab scheduling. The Primary operator is the physician who usually stands nearest to the C-arm. In most cases in Beaumont this is a Cardiology Fellow in cardiac catheterization cases and Attending Physician for the EP cases. The Secondary operator is the physician who typically stands to the right of the primary operator and in most cases is the attending cardiologist or scrub assistant (nurse/technician). The Nurse or Anesthesia team typically circulates in the room and is responsible for monitoring the patient, administering medications and obtaining equipment for the procedure.

Two methods will be used to measure radiation dose during the catheterization procedure. The Real-time Dosimeter Badge (RaySafe) and the Landauer Luxel Aluminium Oxide Dosimeter Badges. Cardiac Catheterization and electrophysiology implant procedures will be performed according to standard guidelines.

Participants will be randomized 1:1 to either cardiac catheterization without ControlRad or cardiac catheterization with the ControlRad system. The same 1:1 randomization process will be applied to the EP patient population. Participants will be blinded to the randomization.

Once procedure is done,participation also ended and the badges will be removed by the Radiation Safety Officer or research coordinator.

ELIGIBILITY:
Inclusion Criteria:

* - Patient

  * Scheduled to undergo left heart catheterization with angiography, and/or percutaneous coronary intervention
  * Scheduled to undergo pacemaker or ICD implant
  * EP device upgrade
  * Able to provide written informed consent prior to the procedure
  * Age ≥18 years
* Physicians and Staff o Able to provide consent for the study

Exclusion Criteria:

* - Patient

  * Cardiogenic shock
  * Reason for cath procedure is pericardiocentesis
  * Subcutaneous ICDs
  * Lead revisions
  * Inability to provide informed consent
  * Pregnant
* Physicians and Staff

  * Those who are not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Dixon, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ControlRad System | Without ControlRad System
Started | 85 | 85
Completed | 85 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ControlRad System | Without ControlRad System | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (4.6) | 57.1 (9.9) | 63.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 50 | 49 | 99
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Radiation Dose to Primary Operator (RaySafe), Cardiac Catheterization
Description: Median effective radiation dose in microsievert (μSv) to the primary operator at the thyroid. This was measured using a RaySafe dosimeter to assess the radiation dose in each case.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: This outcome measured only the cardiac catheterization procedures, 42 participants in the ControlRad group and 38 in the group without ControlRad
Measure: Median (Inter-Quartile Range); unit: microsievert
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
microsievert | 18 [7 to 35] | 39 [19 to 61]

2. Primary Outcome: Radiation Dose to Primary Operator (Luxel Dosimeter), Cardiac Catheterization
Description: Mean effective radiation dose in microsievert (μSv) to the primary operator at the thyroid. This was measured using a single Luxel dosimeter over all cases to assess the cumulative dose in the study arm.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: This outcome measured only the cardiac catheterization procedures, 42 participants in the ControlRad group and 38 in the group without ControlRad. A single badge was used for all cases, the result is provided as a number per arm. The number is cumulative of the arm with no measure of dispersion.
Measure: Number; unit: microsievert
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
microsievert | 18 | 41

3. Primary Outcome: Radiation Dose to Primary Operator, EP Procedure (Luxel)
Description: Mean effective radiation dose in microsievert (μSv) to the primary operator at the end of each EP implant procedure. A single Luxel dosimeter was and a cumulative dose was recorded.
Time Frame: During each EP implant procedure, an average of 90 minutes
Population: This outcome measured only the EP procedures, 43 in the ControlRad group and 47 in the Without ControlRad group. A single badge was used for all cases, the result is provided as a number per arm. The number is cumulative of the arm with no measure of dispersion.
Measure: Number; unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
microsieverts | 21.7 | 58.1

4. Primary Outcome: Radiation Dose to Primary Operator, EP Procedure (RaySafe)
Description: Median effective radiation dose in microsievert (μSv) to the primary operator at the end of each EP implant procedure using a RaySafe dosimeter. This is measured after each case.
Time Frame: During each EP implant procedure, an average of 90 minutes duration
Population: This outcome measured only the EP procedures, 43 in the ControlRad group and 47 in the Without ControlRad group.
Measure: Median (Inter-Quartile Range); unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
microsieverts | 25 [15 to 69.5] | 61 [25.5 to 149]

5. Secondary Outcome: Radiation Dose to Secondary Operator, Cardiac Catheterization (RaySafe)
Description: Median effective radiation dose (μSv) to the secondary operator at the thyroid. This was measured using a RaySafe dosimeter to assess the radiation dose in each case.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: microsievert
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
microsievert | 12 [6 to 22] | 21 [13 to 49]

6. Secondary Outcome: Radiation Dose to Secondary Operator (Luxel Dosimeter), Cardiac Catheterization
Description: Mean effective radiation dose in microsievert (μSv) to the secondary operator at the thyroid. This was measured using a single Luxel dosimeter over all cases to assess the cumulative dose in the study arm.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: as for outcome 2
Measure: Number; unit: microsievert
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
microsievert | 13 | 26

7. Secondary Outcome: Radiation Dose to Nurse or Anesthetist, Cardiac Catheterization (RaySafe)
Description: Median effective radiation dose in microsievert (μSv) to the Nurse 0r Anesthetist at the thyroid. This was measured using a RaySafe dosimeter to assess the radiation dose in each case.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: microsievert
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
microsievert | NA [NA to NA] — Dosage data unreliable as it is below lower limits of detection | NA [NA to NA] — Dosage data unreliable as it is below lower limits of detection

8. Secondary Outcome: Radiation Dose to Nurse or Anesthetist, Cardiac Catheterization (Luxel)
Description: Mean effective radiation dose in microsievert (μSv) to the Nurse or Anesthetist at the thyroid. This was measured using a single Luxel dosimeter over all cases to assess the cumulative dose in the study arm.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: as for outcome 1
Measure: Number; unit: microsievert
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
microsievert | NA — Dosage data unreliable as it is below lower limits of detection | NA — Dosage data unreliable as it is below lower limits of detection

9. Secondary Outcome: Radiation Dose to Patient, Cardiac Catheterization
Description: Median radiation dose-area product (DAP) to the patient at the end of each cardiac catheterization case using data from a fluoroscopy machine. DAP is defined as the absorbed dose multiplied by the area irradiated micro-gray μGy*m^2.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: μGy*m^2
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
μGy*m^2 | 2276 [1179 to 3321] | 3487 [2257 to 5977]

10. Secondary Outcome: Radiation Dose in Cath Lab Room #5, Cardiac Catheterization
Description: Mean radiation dose microsieverts (μSv) at the end of each cardiac catheterization case at a standard location on the wall of the catheterization laboratory. This was measured using a single Luxel dosimeter over all cases to assess the cumulative dose in the study arm.
Time Frame: During each cardiac catheterization, an average of 90 minutes
Population: as for outcome 2
Measure: Number; unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 42 | 38
microsieverts | 15 | 25

11. Secondary Outcome: Radiation Dose to Secondary Operator, EP Procedure (RaySafe)
Description: Mean effective radiation dose (μSv) to the secondary operator at the at the thyroid. This was measured using a RaySafe dosimeter to assess the radiation dose in each case.
Time Frame: During each EP implant procedure, an average of 90 minutes
Population: This outcome measured only the EP procedures, 43 in the ControlRad group and 47 in the Without ControlRad group.
Measure: Median (Inter-Quartile Range); unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
microsieverts | 3 [1.5 to 5] | 5 [3 to 16]

12. Secondary Outcome: Radiation Dose to Secondary Operator, EP Procedure (Luxel)
Description: Mean effective radiation dose (μSv) to the secondary operator at the at the thyroid. This was measured using a single Luxel dosimeter over all cases to assess the cumulative dose in the study arm.
Time Frame: During each EP implant procedure, an average of 90 minutes
Population: as for outcome 3
Measure: Number; unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
microsieverts | 1.6 | 9

13. Secondary Outcome: Radiation Dose to Nurse or Anesthetist, EP Procedure (RaySafe)
Description: as for outcome 1
Time Frame: During each EP implant procedure, an average of 90 minutes
Population: This outcome measured only the EP procedures, 43 in the ControlRad group and 47 in the Without ControlRad group.
Measure: Median (Inter-Quartile Range); unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
microsieverts | 0 [0 to 2] | 2 [0 to 10]

14. Secondary Outcome: Radiation Dose to Nurse or Anesthetist, EP Procedure (Luxel)
Description: as for outcome 2
Time Frame: During each EP implant procedure, an average of 90 minutes
Population: as for outcome 3
Measure: Number; unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
microsieverts | 0 | 3.8

15. Secondary Outcome: Radiation Dose to Patient, EP Procedure
Description: Mean radiation dose-area product (DAP) to the patient at the end of each EP implant procedure using data from a fluoroscopy machine. DAP is defined as the absorbed dose multiplied by the area irradiated (μGy*m^2)
Time Frame: During each EP implant procedure, an average of 30-45 minutes of active radiation
Population: This outcome measured only the EP procedures, 43 in the ControlRad group and 47 in the Without ControlRad group.
Measure: Median (Inter-Quartile Range); unit: μGy*m^2
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
μGy*m^2 | 43.7 [26 to 95.9] | 72.5 [22.7 to 131.5]

16. Secondary Outcome: Radiation Dose in Cath Lab Room #5, EP Procedure
Description: Mean radiation dose (μSv) at the end of each EP implant procedure at a standard location on the wall of the catheterization laboratory. This was measured using a single Luxel dosimeter over all cases to assess the cumulative dose in the study arm.
Time Frame: During each EP implant procedure, an average of 90 minutes
Population: as for outcome 3
Measure: Number; unit: microsieverts
Arm/Group | ControlRad System | Without ControlRad System
Number analyzed (Participants) | 43 | 47
microsieverts | 0 | 0

ADVERSE EVENTS:
Time Frame: During each cardiac catheterization/EP procedure, an average of 90 minutes
Arm/Group | ControlRad System | Without ControlRad System
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 1/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ControlRad System (N=85) | Without ControlRad System (N=85)
Cardiac Perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04404257/Prot_SAP_000.pdf